CLINICAL TRIAL: NCT02534155
Title: High and Intermediate Risk Degenerative Mitral Regurgitation Treatment: A Randomized Controlled Trial Comparing MitraClip® to Surgical Therapy
Brief Title: High and Intermediate Risk Degenerative Mitral Regurgitation Treatment: A Trial Comparing MitraClip® to Surgical Therapy
Acronym: HiRiDe
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HiRiDe
Record Dates: First submitted 2015-08-06; First posted 2015-08-27 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Mitral Valve Insufficiency
Keywords: MitraClip®; MR; DMR; high-risk patients; mitral regurgitation; surgery; intermediate risk patients
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MitraClip® Therapy (Active Comparator): MitraClip® system is a CE marked medical device, which consists of two parts (Clip Delivery System and Steerable Guide Catheter). It is a single sized, percutaneously implanted mechanical Clip. The MitraClip® device grasps and coapts the mitral valve leaflets resulting in fixed approximation of the mitral leaflets throughout the cardiac cycle. The procedure is performed in the cardiac catheterisation laboratory with echocardiographic and fluoroscopic guidance while the patient is under general anaesthesia.
  Interventions: Device: MitraClip®
- Surgery (Active Comparator): Surgical therapy of degenerative mitral regurgitation: repair or replacement of mitral valve, clinical standard
  Interventions: Procedure: Mitral valve Surgery

INTERVENTIONS:
Device: MitraClip® — one or more (if needed) MitraClip® devices are placed on the leaflets of the mitral valve during catheterisation in a catheter laboratory
  Arms: MitraClip® Therapy
Procedure: Mitral valve Surgery — Repair or replace mitral valve
  Arms: Surgery

SUMMARY:
The study is comparing MitraClip® to Surgical therapy in high and intermediate risk patients, who should be older than 18 years, and shall evaluate safety and efficacy of MitraClip® vs. surgery in high or intermediate risk patients. The patients will be randomised (MitraClip® or Surgery). The Study Follow-Up includes 4 visits after procedure (hospital discharge, 1, 6, 12 months post-procedure).

DETAILED DESCRIPTION:
Two-arm, multi-centre, randomised prospective study comparing MitraClip® to Surgical therapy in high and intermediate risk patients. Patients should be older than 18 years and high and intermediate risk is defined by a score (for MV repair) >= 3% and <= 10% or as determined by the local Heart Team (which should include a surgeon and a cardiologist), based on the evidence that STS risk calculator may not identify all possible risk factors. Patients are selected upon clinical conditions and severity of MR. Anatomical feasibility is assessed by ECHO, according to the IFU (information for use).

The purpose of the trial is to evaluate safety and efficacy of MitraClip® vs. surgery in high and intermediate risk patients with DMR. Study Follow-Up includes the following visits after procedure: Hospital discharge, 1, 6, 12 months post-procedure.

Primary Endpoints are the 30-day safety superiority (ITT analysis) and the 12-month efficacy non-inferiority (ITT analysis) of the MitraClip®. The overall rate of Serious Adverse Events (SAEs) and Serious Adverse Device Events (SADEs) until 12 months and the MR Severity reduction at 6 and 12 month in the MitraClip® and Surgery groups are Secondary Endpoints

ELIGIBILITY:
Inclusion Criteria:

* Gender: Both, male and female
* Minimum Age: 18 Years
* Maximum Age: no maximum age
* Severe (4+) DMR (degenerative mitral regurgitation), or 3+ DMR
* NYHA Functional Class III or IV
* Mitral valve anatomy should be suitable for both MitraClip® and Mitral valve surgery (repair or replacement)
* Subjects meet the following conditions:

Age >18 and high or intermediate risk patients with an STS calculated mortality (using the repair calculator) >=3% and <=10% or as determined by the local Heart Team (which should include a surgeon and a cardiologist), based on the evidence that STS risk calculator may not identify all possible risk factors

* patient is operable
* Signed by the subject and dated approved informed consent prior to any study related procedure
* Available and able to return to study site for post-procedural follow-up examination

Exclusion Criteria:

* Patient incapable to approve the informed consent or Emergency Cases
* functional mitral valve pathology
* evolving endocarditis or active endocarditis in the last 3 months
* heavily calcified leaflets
* subjects in whom transesophageal echocardiography is contraindicated
* subjects in whom transseptal catheterisation is contraindicated
* presence of any known life threatening (non-cardiac major or progressive disease), non-cardiac disease that will limit the subject's life expectancy to less than one year
* currently participating in the study of an investigational drug or device
* untreated clinically significant CAD requiring revascularisation
* any percutaneous coronary, carotid, endovascular intervention or carotid surgery within 30 days or any coronary or endovascular surgery within 3 months
* prior mitral valve leaflet surgery or any currently implanted prosthetic mitral valve, or any prior transcatheter mitral valve procedure
* concomitant and significant aortic or tricuspid valve pathology
* CVA or TIA within 6 months or severe carotid stenosis (>70% assessed by Ultrasound)
* contraindication or known allergy to device's components, aspirin, anti-coagulation therapy or contrast media that cannot be adequately managed with premedication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
30-day safety superiority (ITT analysis): Major Adverse Event Composite | 30 days
  The study is powered to show superiority for safety of an endovascular treatment strategy with the MitraClip® as compared to a surgical treatment strategy. The primary safety endpoint is a Major Adverse Event Composite (MAE) including all-cause death, prolonged ventilation (>48h), renal failure, stroke and need for non-elective cardiovascular or thoracic surgery (defined as any kind of cardiovascular and thoracic surgery performed within 30 days from the index procedure and non anticipated prior to the procedure). The analysis of the primary safety endpoint is a test of superiority for the proportion of subjects free from the composite of safety events in the Device vs. the Surgery group at 30 days.
12-month efficacy non-inferiority (ITT analysis): Proportion of responders in the Device vs. the Surgery group | 12 month
  The study is powered to show non-inferiority for clinical efficacy of an endovascular treatment strategy with the MitraClip® as compared to a surgical treatment strategy. The primary effectiveness endpoint is a test of non-inferiority for the proportion of responders in the Device vs. the Surgery group at 12 months. Patients are defined as responders if they are alive with at least a 1-grade improvement in NYHA Functional Class at 12 months over baseline and have not experienced a HF hospitalization within 12 months of randomization (MitraClip® procedure or Surgery).

SECONDARY OUTCOMES:
Overall rate of Serious Adverse Events (SAEs) and Serious Adverse Device Effects (SADEs) within 12 month | 12 month
  Evaluation of all SAEs and SADEs that occur during the trial
MR Severity reduction at 6 and 12 month | between 6 and 12 month
  MR (Mitral Regurgitation) Severity reduction at 6 and 12 months in the MitraClip® and Surgery groups
NYHA class changes at 6 and 12 months | between 6 and 12 month
  NYHA class changes at 6 and 12 months in the MitraClip® and Surgery groups
Change in 6MWT in 6 and 12 month | between 6 and 12 months
  Change in 6MWT (6 Minute Walking Test) in 6 and 12 months in the MitraClip® and Surgery groups
Change in Quality of Life in 6 and 12 months | between 1 and 12 months
  Change in Quality of Life (MLWHF) at 1,6 and 12 month in the MitraClip® and Surgery groups
Heart failure hospitalisation rate | during 12 months post procedure
  Heart failure hospitalisation rate in the post randomisation in the MitraClip® and Surgery groups
Days alive and out of hospital | during 12 months post procedure
  Days alive and out of hospital in the 12 months post-randomisation in the MitraClip® and Surgery groups
Hospital resources utilisations | during 12 months post procedure
  Hospital resources utillizations: length of stay post-procedure, ICU beds occupancy, need for rehabilitation services
Change in Quality of Life (SF36) in 6 and 12 months | between 1 and 12 months
  Change in SF36 at 1,6 and 12 month in the MitraClip® and Surgery groups

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Maisano, Prof., Principal Investigator — Universitätspital Zürich
Locations (12):
- Germany (6):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Herzzentrum, Cologne
  - Asklepios Klinik Hamburg St. Georg, Hamburg
  - Universitäres Herzzentrum Hamburg GmbH, Hamburg
  - Klinikum der Universität München Großhadern, München
  - Helios Klinikum Siegburg, Siegburg
- Italy (3):
  - Presidio Ospedaliero Ferrarotto Alessi, Catania
  - San Raffaele Hospital, Milan
  - Policlinico Tor Vergata, Roma
- Switzerland (3):
  - Universitätsspital Zürich, Zurich, Canton of Zurich
  - Inselspital Bern, Bern
  - Fondazione Cardiocentro Ticino, Lugano